CLINICAL TRIAL: NCT05301166
Title: THE EFFICIENCY OF TECHNOLOGY-BASED MOTIVATION EDUCATION MADE ACCORDING TO THE HEALTH BELIEF MODEL ON OBESITY UNIVERSITY STUDENTS' BELİEFS AND ATTITUDES, NUTRITION-EXERCISE BEHAVIORS, SELF-EFFICIENCY AND WEIGHT MANAGEMENT.
Brief Title: THE EFFICIENCY OF TECHNOLOGY-BASED MOTIVATION EDUCATION ON OBESITY UNIVERSITY STUDENTS' WEIGHT MANAGEMENT.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, MUHAMMED AKİF SAMİ TOKER, Research Assistant, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TBMEP-MAST-01
Record Dates: First submitted 2022-03-19; First posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Overweight and Obesity
Keywords: Obesity; Motivational Interviewing; Health Belief Model; Nursing
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Quasi-experimental pretest-posttest randomized controlled trial.
Who Masked: Outcomes Assessor
Masking Description: In the randomized controlled study, blinding will be done in terms of statistician and reporting. The data regarding the pre-test and post-tests will be collected by another researcher who does not know who is in the experimental and control group, and the research data will be coded and transferred to the computer environment by another researcher without specifying the experimental and control groups. The analysis of the data coded in terms of groups will be done by a statistics expert. After the statistical analyzes are made and the research report is written, the assistant researcher will explain the coding for the experimental and control groups. In this way, a single blinding application was planned for the researcher.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Group (Experimental): The intervention group of the RCT consisted of 42 randomly selected students with a Body Mass Index (BMI) score of 25 and above, who were evaluated by inclusion and exclusion criteria.
  Students in the intervention group will participate in the Technology-Based Motivation Education Program. This program will last 4 months.
  * Students in the intervention group will conduct semi-structured individual motivational interviews, consisting of 6 sessions in total, prepared according to the components of the Health Belief Model.
  * Students in the intervention group will access the web-based education and motivation program that supports motivational interviews by logging into the website prepared for the study.
  Interventions: Behavioral: Technology Based Motivation Education Program
- Control Group (Other): The intervention group of the RCT consisted of 42 randomly selected students with a Body Mass Index (BMI) score of 25 and above, who were evaluated by inclusion and exclusion criteria.
  * Students in the control group will only participate in the web-based education of the Technology-Based Motivation Education Program prepared according to the Health Belief Model for obesity.
  * Students in the control group will be given face-to-face or online interviews once a month for 4 months, lasting 10-15 minutes, in accordance with the web-based education content.
  Interventions: Other: Web Based Education

INTERVENTIONS:
Behavioral: Technology Based Motivation Education Program — Technology-Based Motivation Education Program consists of web-based education, motivation program and individual motivation interviews. This program will be prepared according to the Health Belief Model (HBM). It will be applied for 4 months. Participants will take a pre-test before starting the program and a post-test at the end of the program. Individual motivation interviews will be 6 sessions in total. A website will be prepared for the Technology Based Motivation Education Program. This website consists of two parts, a web-based education and motivation program for obesity. The motivation program will enable the participant to follow the program and receive motivational messages.
  Arms: Interventional Group
Other: Web Based Education — Students in the control group will participate in web-based educations on obesity prepared only according to the Health Belief Model in the Technology-Based Motivation Education Program. Individual interviews supporting web-based education will be held with the control group once a month.
  Arms: Control Group

SUMMARY:
The aim of this study is to determine the effects of technology-based motivation education prepared according to the health belief model on obesity-related beliefs and attitudes, nutrition-exercise behaviors, self-efficacy and weight management in obese university students.

DETAILED DESCRIPTION:
It is stated that the university period is risky in terms of acquiring negative health behaviors that may cause overweight and obesity. In addition, it is emphasized that the transition from overweight to obesity usually occurs between the ages of 18-29. There are non-formal education programs on obesity management for adolescence and adulthood. It is noteworthy that young people in the university period are not adequately represented in the current education programs, and at the same time, education programs specific to young people are limited. The aim of this study is to determine the effects of technology-based motivation education prepared according to the health belief model on obesity-related beliefs and attitudes, nutrition-exercise behaviors, self-efficacy and weight management in obese university students. This quasi-experimental pretest-posttest randomized controlled study will be carried out at Sivas Cumhuriyet University Suşehri Health College and Suşehri Timur Karabal Vocational School between February 1, 2022 and September 15, 2022. The sample of the study will consist of 84 students (experimental group n= 42 and control group n=42). A web-based technology based motivation program including motivational interviewing will be applied to the students in the experimental group. The control group will only receive web-based education on obesity. Data will be collected using Personal Information Form, Obesity Health Belief Model Scale, Nutrition-Exercise Behavior Scale, Self-Efficacy-Efficacy Scale and Website Usability Scale. physical measurements; A digital height-weight meter will be used for BMI measurement, and a tape measure will be used for waist and hip circumference. Whether the data is normal or not will be determined by Kolmogorov-Smirnov, Shapiro Wilk tests. In order to determine whether there is a difference in the research, necessary parametric and nonparametric tests will be used depending on whether the assumptions are met or any or all of the assumptions are not met.

ELIGIBILITY:
Inclusion Criteria:

* 18-25 age range
* Body Mass Index (BMI) ≥ 25.0,
* Having internet access with a computer, tablet or mobile device.

Exclusion Criteria:

* Under 18 years old or over 25 years old,
* BMI < 25.0,
* Continuously using regular medication,
* Presence of a pre-existing health problem (having a surgical operation in the last three months, having diseases with metabolic syndrome, being diagnosed with cancer, being diagnosed with an eating disorder, being diagnosed with a psychological illness, and being physically disabled),
* Participating in any weight management program in the last three months,
* Pregnancy.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-07-15 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Obesity Health Belief Model Scale | 4 Months
  The scale assesses individuals' beliefs and attitudes towards weight loss. It consists of 32 items in total. The scale has five sub-dimensions that can be used independently of each other: importance of health, sensitivity, seriousness, perception of benefit and disability. The cronbach alpha coefficient of the scale is 0.80.
Nutrition-Exercise Behavior Scale | 4 Months
  The scale was developed to identify feeding-related behaviors. It consists of 45 items. The scale has four sub-dimensions: psychological (addicted) eating behavior, healthy diet-exercise behavior, unhealthy diet-exercise behavior, and meal order. The Cronbach Alpha reliability coefficient of the scale is 0.85.
Self-Effectiveness-Efficacy Scale | 4 Months
  The scale measures the perception of general self-efficacy-effectiveness that is not specific to any field. The scale consists of 23 items. The scale has four sub-dimensions: initiating the behavior, maintaining the behavior, completing the behavior and struggling with obstacles. The cronbach alpha coefficient of the Turkish version of the scale is 0.81.

CONTACTS AND LOCATIONS:
Overall Officials: Nuran GÜLER, Prof. Dr., Study Director — Cumhuriyet University
Locations (1):
- Sivas Cumhuriyet University, Sivas, Turkey (Türkiye)